CLINICAL TRIAL: NCT02268604
Title: Safety, Pharmacodynamics, and Pharmacokinetics After Multiple Oral Doses of 200 and 300 mg BIIB 722 CL Tablet Tid and 300 and 450 mg BIIB 722 CL Tablet Bid Over 7 Days to Healthy Volunteer Subjects. An Open Study, Placebo-controlled Randomised Double Blind at Each Dose Level.
Brief Title: Safety, Pharmacodynamics, and Pharmacokinetics After Multiple Different Oral Doses of BIIB 722 CL Tablets in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1180.2
Record Dates: First submitted 2014-08-21; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIIB 722 CL (Experimental)
  Interventions: Drug: BIIB 722 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB 722 CL
  Arms: BIIB 722 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess safety, pharmacodynamics and pharmacokinetics of BIIB 722 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* 18 to 55 years of age
* Broca index >= -20% and <= +20%
* Written informed consent according to Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs, which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration of during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma (AUC) | up to day 7
Maximum measured concentration of the analyte in plasma (Cmax) | up to day 7
Time to maximum measured concentration of the analyte in plasma (tmax) | up to day 7
Total mean residence time of the analyte in the body (MRTtot) | up to day 7
Total clearance of the analyte in plasma (CLtot/f) | up to day 7
Terminal half-life of the analyte in plasma (t1/2) | up to day 7
Amount of the analyte excreted in urine (Ae) | up to day 7
Dose proportionality | up to day 7
  assessed by AUC
Accumulation factor | up to day 7
  (predose concentration/concentration after 8 hours)
Time to reach steady state | up to day 7
Thrombocytic Na-H exchange (NHE-1) inhibition by AUC of pH recovery | up to day 7
  in vitro fluorescence

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to day 12
Number of subjects with clinically significant findings in vital functions | up to day 12
Number of subjects with clinically significant findings in laboratory tests | up to day 12